CLINICAL TRIAL: NCT06092658
Title: Cohort Study of Chronic Heart Failure
Status: Completed | Type: Observational
Sponsor: Xiang Xie (Other)
Responsible Party: Sponsor-Investigator, Xiang Xie, professor, Xinjiang Medical University
Organization: Xinjiang Medical University (Other)
Other Study IDs: 202207-019
Record Dates: First submitted 2023-08-21; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Analyze Etiology, Comorbidities, Clinical Characteristics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No Intervention: No Intervention
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — no intervention

SUMMARY:
The purpose is to understand the clinical characteristics of chronic heart failure as soon as possible, analyze the etiology, comorbidities, clinical characteristics, and treatment of heart failure patients, observe the gap between real-world clinical practice and guideline recommendations, and provide reference for the improvement of heart failure prevention and treatment in China.

DETAILED DESCRIPTION:
Inclusion criteria:

1. Accompanied by difficulty breathing, fatigue, or decreased activity tolerance;
2. Signs of fluid retention (pulmonary congestion and peripheral edema);
3. Echocardiography shows abnormalities in cardiac structure and/or function;
4. Elevated levels of natriuretic peptide: B-type natriuretic peptide (BNP)>35 ng/L and/or N-terminal B-type proBNP (NT proBNP)>125 ng/L.
5. HF hospitalization recorded within the previous 12 months

Exclusion criteria:

1. Concomitant severe liver function, renal failure, or other severe system dysfunction
2. Poor compliance, inability to obtain information, or voluntary refusal to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Accompanied by difficulty breathing, fatigue, or decreased activity tolerance;
2. Signs of fluid retention (pulmonary congestion and peripheral edema);
3. Echocardiography shows abnormalities in cardiac structure and/or function;
4. Elevated levels of natriuretic peptide: B-type natriuretic peptide (BNP)>35 ng/L and/or N-terminal B-type proBNP (NT proBNP)>125 ng/L.

Exclusion Criteria:

1. Concomitant severe liver function, renal failure, or other severe system dysfunction
2. Poor compliance, inability to obtain information, or voluntary refusal to participate in this study.

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20000 (Actual)
Dates: Start 2012-11-20 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
echocardiogram | Follow up will be conducted at baseline, 6 months, 12 months, and 36 months
  ejection fraction,Consider heart failure when the ejection fraction is less than 50%
cardiac marker | Follow up will be conducted at baseline, 6 months, 12 months, and 36 months
  CK，CK-MB，cTnT，cTnI，Mb
serum biochemical indicators | Follow up will be conducted at baseline, 6 months, 12 months, and 36 months
  HDL-cholesterol, mg/dL，LDL-cholesterol, mg/dL，Total cholesterol, mg/dL，Triglycerides, mg/dL

SECONDARY OUTCOMES:
Thyroid Function | Follow up will be conducted at baseline, 6 months, 12 months, and 36 months
  thyroid hormone,Thyroid hormone blood testing: This is the most commonly used method to measure thyroid hormone levels in the blood. Common thyroid hormone indicators include thyroxine, free thyroxine, triiodothyronine, and free triiodothyronine.
Coagulation function indicators | Follow up will be conducted at baseline, 6 months, 12 months, and 36 months
  D-Dimer
Blood routine | Follow up will be conducted at baseline, 6 months, 12 months, and 36 months
  RBC
Blood routine | Follow up will be conducted at baseline, 6 months, 12 months, and 36 months
  WBC
Blood routine | Follow up will be conducted at baseline, 6 months, 12 months, and 36 months
  PLT

IPD SHARING:
Plan to Share IPD: Undecided
undecided